CLINICAL TRIAL: NCT05756738
Title: Acceptance and Feasibility of Hepatitis c Screening Strategies in Social Insertion Centers With Alternative Sentences to Prison and Open System
Brief Title: Acceptance and Feasibility of Hepatitis c Screening Strategies in Social Insertion Centers
Acronym: TGSS_CIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, Principal Investigator, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TGSS_CIS
Record Dates: First submitted 2022-11-20; First posted 2023-03-06 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — Dried Blood Spot Testing

STUDY DESIGN:
Intervention Model Description: A randomized study will be designed in which all persons attending the Social Insertion Center (CIS) to serve alternative sentences to prison will be invited to participate. In order to study the prevalence of these persons compared to persons in open system, the latter will be offered to take the diagnostic test in situ at the CIS premises.
  Persons with alternative sentences to prison will be informed of the study and, according to the randomization code, will be: a) given an envelope with all the necessary material to carry out the test at home and send it to the hospital for processing or, b) be tested on site at the CIS premises, who will also send it to the hospital for processing by the Central Laboratory of the University Hospital of the Canary Islands.
  All patients who have participated will be notified by telephone of the test result, and patients with a diagnosis of active infection will be contacted and given an appointment to be evaluated and treated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative sentences to prison (Experimental): Persons with alternative sentences to prison will be informed of the study and, according to the randomization code, will be: a) given an envelope with all the necessary material to carry out the test at home and send it to the hospital for processing or, b) be tested on site at the the Social Insertion Center premises, who will also send it to the hospital for processing by the Central Laboratory of the University Hospital of the Canary Islands.
  Interventions: Diagnostic Test: Dried blood spot testing
- Open system (Experimental): They will be offered to take the diagnostic test in situ at the the Social Insertion Center premises.
  Interventions: Diagnostic Test: Dried blood spot testing

INTERVENTIONS:
Diagnostic Test: Dried blood spot testing — To evaluate the efficacy defined as the rate of diagnostic tests against hepatitis C virus (HCV) performed with a dried blood spot test

SUMMARY:
Hepatitis C virus (HCV) infection is one of the leading causes of chronic liver disease worldwide. It is a progressive disease that without treatment leads to the development of cirrhosis in approximately 10-20% of patients. With this study the investigators intend to evaluate the efficacy defined as the rate of HCV diagnostic tests performed within a decentralized diagnostic strategy by means of home self-testing compared to the one performed in situ in the population served in Social Insertion Centers (CIS) with alternative prison sentences, in order to study the prevalence and characteristics associated with HCV infection in this population, which is known to be at risk for this disease, and to offer them treatment and cure.

DETAILED DESCRIPTION:
A randomized study will be designed in which all persons attending the Social Insertion Center to serve alternative sentences to prison will be invited to participate on a voluntary basis, with prior informed consent. In order to study the prevalence of these persons compared to persons in open system, the latter will be offered, with prior informed consent, to take the diagnostic test in situ at the CIS premises. All persons will be given a survey with sociodemographic and clinical variables to identify predictor factors.

People with alternative sentences to prison will be informed of the study and, according to the randomization code, will be: a) given an envelope with all the necessary material to carry out the test at home and send it to the hospital for processing or, b) be tested on site at the CIS premises by the CIS nurse, who will also send it to the hospital for processing within 30 days by the Central Laboratory of the University Hospital of the Canary Islands.

ELIGIBILITY:
Inclusion Criteria:

* All persons attending the Social Insertion Center for the first time with alternative sentences to prison and in open system.
* Signed informed consent.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Minors under 18 years of age and over 79 years of age.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 854 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants in a HCV screening strategy | 1 year
  To evaluate the efficacy defined as the rate of diagnostic tests against hepatitis C virus (HCV) performed within a decentralized diagnostic strategy integrated by self-testing at home compared to that performed in situ in the population served in a Social Insertion Center with alternative prison sentences.

SECONDARY OUTCOMES:
Prevalence of HCV | 1 year
  To study the prevalence and characteristics of patients with active HCV infection who are treated in the Social Insertion Center with alternative prison sentences compared to those in open system, so better and more specialized screening strategies are developed.

CONTACTS AND LOCATIONS:
Overall Officials: Hernández Guerra, Principal Investigator — University of La Laguna
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association for Study of Liver. EASL Clinical Practice Guidelines: management of hepatitis C virus infection. J Hepatol. 2014 Feb;60(2):392-420. doi: 10.1016/j.jhep.2013.11.003. Epub 2013 Dec 9. No abstract available. PMID 24331294
- [Background] Baumert TF, Juhling F, Ono A, Hoshida Y. Hepatitis C-related hepatocellular carcinoma in the era of new generation antivirals. BMC Med. 2017 Mar 14;15(1):52. doi: 10.1186/s12916-017-0815-7. PMID 28288626
- [Background] Westbrook RH, Dusheiko G. Natural history of hepatitis C. J Hepatol. 2014 Nov;61(1 Suppl):S58-68. doi: 10.1016/j.jhep.2014.07.012. Epub 2014 Nov 3. PMID 25443346
- [Background] Buti M, Dominguez-Hernandez R, Casado MA, Sabater E, Esteban R. Healthcare value of implementing hepatitis C screening in the adult general population in Spain. PLoS One. 2018 Nov 28;13(11):e0208036. doi: 10.1371/journal.pone.0208036. eCollection 2018. PMID 30485377
- [Background] Juanbeltz R, Perez-Garcia A, Aguinaga A, Martinez-Baz I, Casado I, Burgui C, Goni-Esarte S, Reparaz J, Zozaya JM, San Miguel R, Ezpeleta C, Castilla J; EIPT-VHC Study Group. Progress in the elimination of hepatitis C virus infection: A population-based cohort study in Spain. PLoS One. 2018 Dec 4;13(12):e0208554. doi: 10.1371/journal.pone.0208554. eCollection 2018. PMID 30513107
- [Background] Morales-Arraez D, Hernandez-Guerra M. Electronic Alerts as a Simple Method for Amplifying the Yield of Hepatitis C Virus Infection Screening and Diagnosis. Am J Gastroenterol. 2020 Jan;115(1):9-12. doi: 10.14309/ajg.0000000000000487. No abstract available. PMID 31833860
- [Background] Crespo J, Albillos A, Buti M, Calleja JL, Garcia-Samaniego J, Hernandez-Guerra M, Serrano T, Turnes J, Acin E, Berenguer J, Berenguer M, Colom J, Fernandez I, Fernandez Rodriguez C, Forns X, Garcia F, Rafael Granados, Lazarus JV, Molero JM, Molina E, Perez Escanilla F, Pineda JA, Rodriguez M, Romero M, Roncero C, Saiz de la Hoya P, Sanchez Antolin G. Elimination of hepatitis C. Positioning document of the Spanish Association for the Study of the Liver (AEEH). Gastroenterol Hepatol. 2019 Nov;42(9):579-592. doi: 10.1016/j.gastrohep.2019.09.002. Epub 2019 Oct 5. English, Spanish. PMID 31594683
- [Background] Bedford J, Enria D, Giesecke J, Heymann DL, Ihekweazu C, Kobinger G, Lane HC, Memish Z, Oh MD, Sall AA, Schuchat A, Ungchusak K, Wieler LH; WHO Strategic and Technical Advisory Group for Infectious Hazards. COVID-19: towards controlling of a pandemic. Lancet. 2020 Mar 28;395(10229):1015-1018. doi: 10.1016/S0140-6736(20)30673-5. Epub 2020 Mar 17. No abstract available. PMID 32197103
- [Background] Morales-Arraez D, Hernandez-Bustabad A, Medina-Alonso MJ, Santiago-Gutierrez LG, Garcia-Gil S, Diaz-Flores F, Perez-Perez V, Nazco J, Fernandez de Rota Martin P, Gutierrez F, Hernandez-Guerra M. Telemedicine and decentralized hepatitis C treatment as a strategy to enhance retention in care among people attending drug treatment centres. Int J Drug Policy. 2021 Aug;94:103235. doi: 10.1016/j.drugpo.2021.103235. Epub 2021 Apr 7. PMID 33838399
- [Background] Saiz de la Hoya P, Marco A, Garcia-Guerrero J, Rivera A; Prevalhep study group. Hepatitis C and B prevalence in Spanish prisons. Eur J Clin Microbiol Infect Dis. 2011 Jul;30(7):857-62. doi: 10.1007/s10096-011-1166-5. Epub 2011 Jan 28. PMID 21274586
- [Background] Sterling RK, Cherian R, Lewis S, Genther K, Driscoll C, Martin K, Goode MB, Matherly S, Siddiqui MS, Luketic VA, Stravitz RT, Puri P, Lee H, Smith P, Patel V, Sanyal AJ. Treatment of HCV in the Department of Corrections in the Era of Oral Medications. J Correct Health Care. 2018 Apr;24(2):127-136. doi: 10.1177/1078345818762591. Epub 2018 Mar 22. PMID 29566611
- [Background] Foschi A, Casana M, Radice A, Ranieri R, d'Arminio Monforte A. Hepatitis C management in prisons: An insight into daily clinical practice in three major Italian correctional houses. Hepatology. 2016 Nov;64(5):1821-1822. doi: 10.1002/hep.28609. Epub 2016 May 31. No abstract available. PMID 27118063
- [Background] Cuadrado A, Cobo C, Mateo M, Blasco AJ, Cabezas J, Llerena S, Fortea JI, Lazaro P, Crespo J. Telemedicine efficiently improves access to hepatitis C management to achieve HCV elimination in the penitentiary setting. Int J Drug Policy. 2021 Feb;88:103031. doi: 10.1016/j.drugpo.2020.103031. Epub 2020 Nov 19. PMID 33221615
- [Background] Crespo J, Llerena S, Cobo C, Cabezas J. Is HCV elimination possible in prison? Rev Esp Sanid Penit. 2017 Dec;19(3):70-73. doi: 10.4321/S1575-06202017000300001. No abstract available. PMID 29364331